CLINICAL TRIAL: NCT05221242
Title: A Randomized Split-mouth Clinical Trial of Partial Laminate Veneers Bonded With Two Different Resin Composite Luting Agents
Brief Title: Clinical Trial on Ceramic Partial Laminate Veneers With Different Luting Agents
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Arturo Prat (Other)
Collaborators: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Gerardo Duran Ojeda, Doctor of Dental Surgery, Universidad Arturo Prat
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-07-10-2021
Record Dates: First submitted 2022-01-10; First posted 2022-02-02 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: partial laminate veneers; sectional veneers; ceramic fragments

STUDY DESIGN:
Intervention Model Description: In this study, two different luting resin cements will be used to bond ceramic partial laminate veneers. This is a randomized split mouth clinical trial, in which only maxillary anterior teeth will be treated with partial veneers (maximum 6 teeth, upper incisors and canines. This zone is called sector 2). For this purpose, sector 2 will be divided in two sides (right and left), and randomization will be performed to select a conventional resin cement or a preheated resin composite luting agent as the material of choice for the right or left side of the mouth to bond ceramic partial laminate veneers for every recruited patient. Number of participants is related to the number of restorations.
Masking Description: two observers will evaluate clinically patient's restorations using the modified USPHS criteria and the FDI criteria. Observers will be blinded to the type of luting agent used for the restoration with ceramic partial laminate veneers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with PLV (Experimental): All patients will receive ceramic partial laminate veneers as treatment. As this is a split mouth design, one side of the mouth will receive partial laminate veneers bonded with a conventional light-curing resin cement and the other side of the mouth with a pre-heated resin composite.
  Interventions: Procedure: Conventional Resin Cement vs Preheated Resin Composite

INTERVENTIONS:
Procedure: Conventional Resin Cement vs Preheated Resin Composite — For this study, variolink esthetic resin cement will be used to bond ceramic partial laminate veneers in one side of the maxillary anterior teeth (left or right upper incisors and canines), while, the other side will receive ceramic partial laminate veneers bonded with a preheated resin composite
  Other Names: Variolink Esthetic (Ivoclar Vivadent, Schaan, Liechtenstein); Enamel Plus HFO (Micerium, Avegno, Italy)

SUMMARY:
Partial laminate veneers is a type of dental restoration made of a glass-matrix ceramic used to restore small teeth fractures, or to correct morphology defects of teeth (i.e.: diastema, conoid teeth or small misalignment). As tooth surface reduction, or tooth preparation is not needed for this type of restoration, it can be considered as a non-tooth preparation minimally invasive procedure.

As non-preparation is required for the restoration with ceramic partial laminate veneers, bonding relies on adhesion between the intaglio surface of the ceramic restoration and the tooth surface, which in most of the cases is enamel. For this purpose, many light-curing resin cement materials are available for bonding procedures. Nowadays, pre-heated resin composites are available as a resin luting material which has been indicated for laminate veneers and partial indirect posterior restorations.

As pre-heated resin composite has not been yet studied for partial laminate veneers, the objective of this randomized split mouth clinical trial, is to evaluate the survival of ceramic partial laminate veneers when bonded with two different resin composite luting agents.

DETAILED DESCRIPTION:
Patients will be recruited starting the 18th of April 2024. Patients willing to enroll in this study must be over 18 years old, capable to read and sign an informed consent, willing to come back to checkups, with periodontal and pulpal health, having anterior teeth with the need of minimal morphology corrections like diastema, conoid teeth or misaligned teeth, and small fractures. Non vital teeth were not excluded. Patients will poor oral hygiene, active caries lesions are excluded.

Pre Operative Procedures. Informed consent will be given first and ask for every patient to sign it. Face and intraoral photographs will be taken. Initial polyvinylsiloxane (PVS) impressions will be performed and sent to the dental laboratory for wax-up from a digital planning analysis. Prophylaxis, new restorations, endodontic treatment and gingival surgery will be performed based on a mock-up made from bis-acrylic material.

Tooth preparation Most cases won't have tooth surface reduction or preparation. Some cases will need smoothening of the sharp angles or enamel irregularities to prevent fractures during restoration try-in. New impression will be performed with PVS impression material to obtain working models for the elaboration of ceramic partial laminate veneers (PLV) One dental technician will elaborate all the PLV according to the manufacturer instructions.

Adhesive luting procedures. Seating, adaptation and form will be checked firt. Try-in pastes will be used to control shade match of the restorations that will be adhesively luted with Variolink Esthetic (conventional light-curing resin cement), while polarized photography of a small amount of polymerized resin composite will be taken for color selection of the preheated resin composite luting agent (Enamel Plus HFO).

Intaglio surfaces of the ceramic restorations protocol:

1. - Application of 9,5% hydrofluoric acid for 120 seconds.
2. - 1 minute of water rinsing. 5 minutes of ultrasonic bath cleaning with distilled water.
3. - Silane application
4. - Bonding Application (without light-curing):

   * Optibond Fl adhesive for ceramics that will be bonded with Enamel Plus HFO.
5. - Charge of resin cement (without light-curing)

   * Variolink esthetic according to color try-in.
   * Enamel Plus HFO will be pre heated in a resin heater at 69ºC.
6. - Store the restorations of light exposure.

Surface treatment of enamel and dentin (if dentin is exposed):

1. - Apply phosphoric acid for 15 seconds in enamel.
2. - rinse profusely with water for 30 seconds.
3. - air-dry
4. - apply adhesive on tooth surface.
5. - No light-curing.

Restorations will be seated with small finger pressure, excesses of resin cement will be eliminated using brushes. Light-curing will be then performed using soft mode of approximately 650mw/cm2 during 3-5 seconds. A final light-curing in high mode will be performed after 3-5 minutes of waiting at approximately 1200 mw/cm2.

Polishing procedure All restorations will be polished with 2-step diamond spiral wheels under water irrigation.

Evaluation 2 blind observers to the luting procedure performed will evaluate clinically the restorations using the modified USPHS criteria and the FDI (World Dental Federation) criteria for the evaluation of direct and indirect restorations. Also an Impact in Oral Health questionary will be applied to determine the esthetic perception of the applied treatment.

modified USPHS criteria and FDI criteria will be applied at baseline after luting the restorations and every 6 months until a completion of minimum of 24 months.

Impact in Oral Health questionary will be applied at baseline and 6 months after the treatment.

Scanning Electron Microscopy evaluation Every case will receive final impressions immediately after the treatment, and after 24 months to evaluate marginal adaptation under Scanning electron microscopy. Fractography Analysis will be performed of every failure or fracture of the restoration.

Statistical analysis Survival will be measure in percentages. Differences will be measure between baseline and final control.

Kaplan-Meier curves will be used to measure cumulative survival, and log rank (Mantel-Cox) to determine differences between the two groups (bonded with conventional resin cement vs pre heated resin composite)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients able to read and sign an informed consent.
* Patients willing to come back to check-ups.
* Patients without active caries lesions or periodontal disease.
* Patients that need to restore their anterior maxillary teeth (upper incisors or canines) due to small fractures, misaligned teeth, conoid teeth or diastema.
* Non-vital teeth will also be included.

Exclusion Criteria:

* Patients with active caries lesions or periodontal disease.
* Patients with occlusal disfunction or uncontrolled parafunctional habits.
* Patients unwilling to come back to checkups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival Data of Partial Laminate Veneers bonded with Conventional Resin Cement and Preheated Resin Composite | after 36 months
  Survival data will be measured in percentages (0-100%) over the years. Kaplan - Meier curves are used to determine the moment of failure (date, months) Mantel - Cox test will be used to determine differences between the two groups

OTHER OUTCOMES:
Success Data of Partial Laminate Veneers bonded with Conventional Resin Cement and Preheated Resin Composite | after 36 months
  Success will be clinically evaluated using the modified USPHS criteria and the FDI criteria. This criteria are used to evaluate the need of refurbishment, repair or replacement of a restoration using different categories. Scores in FDI criteria range from 1-5 with 1-3 acceptable, 4 un-acceptable but repairable and 5 need for repair.
Assessment of Oral Health Impact Profile | after 12 months
  Final outcome with Partial veneers will be measured using the Oral Health Impact Profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Áurea Iquique, Iquique, Chile

IPD SHARING:
Plan to Share IPD: No
The information of patients will be private and not shared. Only researchers included in the Study will be authorized to access patient's data.
  Blind observers won't be able to access patients data to reduce bias.

REFERENCES:
- [Background] Gresnigt MM, Kalk W, Ozcan M. Randomized controlled split-mouth clinical trial of direct laminate veneers with two micro-hybrid resin composites. J Dent. 2012 Sep;40(9):766-75. doi: 10.1016/j.jdent.2012.05.010. Epub 2012 Jun 2. PMID 22664565
- [Background] Sinhori BS, Monteiro S Jr, Bernardon JK, Baratieri LN. CAD/CAM ceramic fragments in anterior teeth: A clinical report. J Esthet Restor Dent. 2018 Mar;30(2):96-100. doi: 10.1111/jerd.12342. Epub 2017 Sep 28. PMID 28960775
- [Background] Gresnigt MMM, Sugii MM, Johanns KBFW, van der Made SAM. Comparison of conventional ceramic laminate veneers, partial laminate veneers and direct composite resin restorations in fracture strength after aging. J Mech Behav Biomed Mater. 2021 Feb;114:104172. doi: 10.1016/j.jmbbm.2020.104172. Epub 2020 Nov 4. PMID 33172798
- [Background] Ceinos R, Pouyssegur V, Allard Y, Bertrand MF. Esthetic rehabilitation of the smile with partial laminate veneers in an older adult. Clin Case Rep. 2018 Jun 4;6(8):1407-1411. doi: 10.1002/ccr3.1593. eCollection 2018 Aug. PMID 30147872
- [Background] Elter B, Aladag A, Comlekoglu ME, Dundar Comlekoglu M, Kesercioglu AI. Colour stability of sectional laminate veneers: A laboratory study. Aust Dent J. 2021 Sep;66(3):314-323. doi: 10.1111/adj.12837. Epub 2021 Apr 7. PMID 33721347
- [Background] Signore A, Kaitsas V, Tonoli A, Angiero F, Silvestrini-Biavati A, Benedicenti S. Sectional porcelain veneers for a maxillary midline diastema closure: a case report. Quintessence Int. 2013 Mar;44(3):201-6. doi: 10.3290/j.qi.a29058. PMID 23444201
- [Background] Gresnigt M, Ozcan M. Esthetic rehabilitation of anterior teeth with porcelain laminates and sectional veneers. J Can Dent Assoc. 2011;77:b143. PMID 22067068
- [Background] Farias-Neto A, Gomes EM, Sanchez-Ayala A, Sanchez-Ayala A, Vilanova LS. Esthetic Rehabilitation of the Smile with No-Prep Porcelain Laminates and Partial Veneers. Case Rep Dent. 2015;2015:452765. doi: 10.1155/2015/452765. Epub 2015 Oct 18. PMID 26568893
- [Background] Horvath S, Schulz CP. Minimally invasive restoration of a maxillary central incisor with a partial veneer. Eur J Esthet Dent. 2012 Spring;7(1):6-16. PMID 22319761